CLINICAL TRIAL: NCT05071287
Title: Precision Metabolic Mechanisms of Low Carbohydrate and Ketogenic Diet
Brief Title: Metabolism of Low Carbohydrate and Ketogenic Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC20190528H
Record Dates: First submitted 2021-08-24; First posted 2021-10-08 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Kidney Disease; Cognitive Function; Weight Loss; Diabetic Control; Type2 Diabetes
Keywords: Weight loss; Healthy lifestyle intervention; Type 2 Diabetes; Renal function
MeSH Terms: conditions — Diabetic Nephropathies; Weight Loss; Diabetes Mellitus, Type 2 | interventions — Telemedicine; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 arms. Randomization will be done in clusters:
  1. overweight/obese adults with type 2 diabetes (T2D) but no chronic kidney disease (CKD)
  2. overweight/obese with T2D without CKD
  3. overweight/obese with early stage CKD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (mHealth+low-fat diet group) (Placebo Comparator): The low-fat group will be asked to restrict total calorie and total fat consumption according to the Look AHEAD intervention and MyPlate guidelines, with 26-44% carbs, 10-30% protein, and less than 30% fat.
  Interventions: Other: mHealth + low-fat diet
- Intervention Group (mHealth + low-carbohydrate/ketogenic diet group) (Experimental): Total calories will be set according to Look AHEAD intervention, and carbohydrate consumption restriction will be set based on recommendations from American Diabetic Association, National Kidney Foundation, and other evidence-based resources. Participants in this group will be asked to consume a low-carb/ketogenic diet. Specially, participants will receive a carbohydrate, protein, and fat intake goal based on 1.5 : 1 ratio (1.5 grams of fat to 1 gram of carbohydrate and protein combined). Daily macronutrient and calorie consumption will be individualized for each participant using ideal body weight as inferred from wrist circumference and activity level. Carbohydrate consumption will be less than 10% (20~50 g), protein 10-20% (1.0~1.2g/kg ideal body weight), and fat 70-80% of total daily energy, respectively. Nutritional ketosis will be reached by consuming such diet (0.5 mmol/L).
  Interventions: Other: mHealth + low-carb/ketogenic diet

INTERVENTIONS:
Other: mHealth + low-fat diet — A restricted total calorie and reduced total fat consumption.
  Arms: Control Group (mHealth+low-fat diet group)
Other: mHealth + low-carb/ketogenic diet — A low-carb/ketogenic diet
  Arms: Intervention Group (mHealth + low-carbohydrate/ketogenic diet group)

SUMMARY:
This study will assess the preliminary efficacy of a lifestyle intervention including low-carb/ketogenic diet and exercise, enhanced by self-monitoring through health technologies on weight and diabetes outcomes (Glucose, HbA1c) and diabetic complications (cognitive function, and renal function) in a 6-month randomized clinical trial in 60 overweight/obese adults with or without T2D. Renal function will be assessed via both traditional and novel biomarkers, including novel metabolites and mitochondrial function.

DETAILED DESCRIPTION:
Participants in both groups will receive standardized health education sessions including lifestyle management, blood glucose control, blood pressure control, and prevention of diabetic complications from trained providers who are also investigators of this study. The lifestyle intervention from the evidence-based Group Lifestyle Balance (GLB) program (http://www.diabetesprevention.pitt.edu/index.php/for-the-public/for-health-providers/group-lifestyle-balance-curriculum/) and Look AHEAD intervention (https://www.lookaheadtrial.org) will be modified for this study. Goal for weight loss and physical activity will be set for each participant based on recommendations from GLB and Look AHEAD. Lifestyle intervention will be delivered through interactive digital lessons. Smart phone and mobile health devices will be used for each participant to self-monitor diet, physical activity, weight, glucose level, blood pressure, and blood ketone (if randomized to the low-car/ketogenic diet group).

Control group (mHealth+ low-fat diet group):

The low-fat group will be asked to restrict total calorie and total fat consumption according to the Look AHEAD intervention and MyPlate guidelines, with 26-44% carbs, 10-30% protein, and less than 30% fat.

Intervention group (mHealth+ low-carb/ketogenic diet group):

The low-carb/ketogenic diet group, will have total calorie set according to Look AHEAD intervention, and carb consumption restriction will be set based on recommendations from American Diabetic Association, National Kidney Foundation, and other evidence-based resources. Participants in this group will be asked to consume a low-carb/ketogenic diet. Specially, participants will receive a carbohydrate, protein, and fat intake goal based on 1.5 : 1 ratio (1.5 grams of fat to 1 gram of carbohydrate and protein combined). Daily macronutrient and calorie consumption will be individualized for each participant using ideal body weight as inferred from wrist circumference and activity level. Carbohydrate consumption will be less than 10% (20~50 g), protein 10-20% (1.0~1.2g/kg ideal body weight), and fat 70-80% of total daily energy, respectively. Nutritional ketosis will be reached by consuming such diet (0.5 mmol/L).

All diet intervention materials will be developed by a registered dietitian according to the evidence-based guidelines. The dietitian will also be responsible to any study activities relevant to diet. These activities include but are not limited to responding to some specific diet questions to study participants and health related measurements relevant to diet changes.

An interventionist, under supervision of a registered dietitian, will interact with each participant from both groups at the beginning of the intervention as an introduction visit, and three individual intervention sessions at month 1, 3, and 5. During the introduction visit, the interventionist will set up a personalized weight loss goal and caloric intake goal with the participants. The individual intervention sessions at month 1, 3 and 5 will be arranged to solve the encountered problems regarding diet, weight loss, caloric intake and action planning.

Additional communication through phone call will be used to support patient dietary changes throughout the study based on their self-monitoring information.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study
2. being 18 and over
3. For overweight/obese adults (BMI≥25kg/m2)

   1. without self-reported diagnosis of Type 2 Diabetes (T2D) or Chronic Kidney Disease (CKD): Estimated Glomerular Filtration Rate (eGFR)≥90mL/min/1.73m2 and urine albumin to creatinine ratio (ACR)<30mg/g within the past 12 months
   2. with Type 2 Diabetes (T2D) but without Chronic Kidney Disease (CKD): Estimated glomerular filtration rate (eGFR)≥90mL/min/1.73m2 and Albumin-to-Creatinine ratio (ACR)<30mg/g within the past 12 months
   3. with early stage Chronic Kidney Disease (CKD): 60≤eGFR<90mL/min/1.73m2 or 30mg/g ≤ACR< 1000mg/g within the 12 months
4. can speak and understand English
5. own a smart phone or tablet that has reliable internet/data access
6. agree to comply with all study requirements

Exclusion Criteria:

1. Patients with triglyceride ≥ 500 mg/dL or with Low-Density Lipoprotein Cholesterol≥ 129mg/dL
2. type 1 diabetes (by self-report)
3. severe psychiatric disorders deemed by investigators, which might interfere with study procedures (by self-report)
4. severe chronic conditions (e.g. severe heart disease, renal disease, cognitive impairment, etc.) that would preclude them from participating
5. unwillingness to sign the consent form and be randomized into a study group
6. enrollment in other low carb/keto diet or weight loss programs
7. inability to walk without assistance (by self-report)
8. under SGLT2 inhibitor treatment
9. being pregnant or breast feeding (by self-report)
10. having plans to leave the city or USA for over 2 weeks within 6 months at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline to 6 months
  Measure of weight change that occurred while assigned to the diet

SECONDARY OUTCOMES:
BMI | Baseline to 6 months
  BMI (Body Mass Index) is a numerical value derived from a person's weight and height, used as a screening tool to classify individuals into weight categories. It is calculated using weight (kg) divided by height (m)2.
HbA1c | Baseline to 6 months
  HbA1c (Hemoglobin A1c) is a blood test that measures the average blood glucose levels over the past 2 to 3 months.
Blood pressure | Baseline to 6 months
  Blood Pressure (BP) is the force exerted by circulating blood against the walls of the arteries. It is measured in millimeters of mercury (mmHg) and recorded as two values: Systolic Pressure and Diastolic Pressure.
Blood lipids | Baseline to 6 months
  Blood lipids refer to the fatty substances found in the bloodstream, including cholesterol and triglycerides.
Estimated Glomerular Filtration rate (eGFR) | Baseline to 6 months
  Measure of change in eGFR in a blood sample.
Albumin-to-Creatinine ratio (ACR) | Baseline to 6 months
  Measure of the change in ACR in urine.
Metabolites | Baseline to 6 months
  Metabolites are small molecules that are intermediates or end products of metabolism.
Mitochondrial DNA | Baseline to 6 months
  Measure of change of mitochondrial function using blood and urine levels

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Baseline to 6 months
  A one page, 30-point test administered to test cognition. MoCA scores range between 0 and 30. A score of 26 or over is considered to have no cognitive impairment, while lower scores imply more cognitive impairment. Tasks include short term memory recall, visuospatial ability tests, attention, concentration and working memory evaluation and language skills.
Gut Metabolomics | Baseline to 6 months
  Measure of changes of gut metabolites using mass spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Du, PhD MPH RN, Principal Investigator — University of Texas Health San Antonio
Locations (2):
- United States (2):
  - University Health System Texas Diabetic Institute, San Antonio, Texas
  - UT Health San Antonio School of Nursing, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The plan to make Individual Participant Data (IPD) available to other researchers has not been decided.

REFERENCES:
- [Derived] Li S, Du Y, Miao H, Sharma K, Li C, Yin Z, Brimhall B, Wang J. Understanding Heterogeneity in Individual Responses to Digital Lifestyle Intervention Through Self-Monitoring Adherence Trajectories in Adults With Overweight or Obesity: Secondary Analysis of a 6-Month Randomized Controlled Trial. J Med Internet Res. 2024 Mar 20;26:e53294. doi: 10.2196/53294. PMID 38506903
- [Derived] Li S, Du Y, Meireles C, Song D, Sharma K, Yin Z, Brimhall B, Wang J. Decoding Heterogeneity in Data-Driven Self-Monitoring Adherence Trajectories in Digital Lifestyle Interventions for Weight Loss: A Qualitative Study. Res Sq [Preprint]. 2024 Jan 19:rs.3.rs-3854650. doi: 10.21203/rs.3.rs-3854650/v1. PMID 38313251